CLINICAL TRIAL: NCT07321626
Title: Efficacy and Safety of Romiplostim N01 in Promoting Platelet Reconstruction After Haploidentical Allogeneic Stem Cell Transplantation in Patients With Hematologic Malignancies
Brief Title: Romiplostim N01 for Platelet Recovery After Haploidentical HSCT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJU-HSCT-ROMN01
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; MDS (Myelodysplastic Syndrome); Delayed Platelet Engraftment; HSCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romiplostim N01 Treatment Arm (Experimental)
  Interventions: Drug: Romiplostim N01; Other: Standard Supportive Care
- Standard Care Control Arm (Active Comparator)
  Interventions: Other: Standard Supportive Care

INTERVENTIONS:
Drug: Romiplostim N01 — Romiplostim N01 is a thrombopoietin receptor agonist (TPO-RA) administered subcutaneously once weekly to promote platelet recovery after haploidentical allogeneic hematopoietic stem cell transplantation (haplo-HSCT). The starting dose is 5 µg/kg, adjusted up to 10 µg/kg according to platelet response. Treatment continues for up to 4 weeks or until platelet counts reach ≥100 × 10⁹/L without transfusion. Standard post-transplant supportive care is provided to all participants.
  Arms: Romiplostim N01 Treatment Arm
Other: Standard Supportive Care — Participants in the control arm will receive standard post-transplant supportive care, including transfusions, growth factors (G-CSF, ESA), and infection prophylaxis as clinically indicated, but will not receive Romiplostim or any other thrombopoietin receptor agonist.

SUMMARY:
This is a prospective, randomized, controlled clinical study designed to evaluate the efficacy and safety of Romiplostim N01 in promoting platelet engraftment after haploidentical allogeneic hematopoietic stem cell transplantation (haplo-HSCT) in patients with hematologic malignancies.

A total of 130 patients who undergo haplo-HSCT for acute myeloid leukemia (AML), myelodysplastic syndromes (MDS), or other hematologic malignancies will be enrolled and randomized 1:1 into a treatment group and a control group. The treatment group will receive Romiplostim N01 subcutaneously once weekly at a starting dose of 5 µg/kg, with dose adjustments based on platelet counts (maximum 10 µg/kg), for up to 4 weeks or until platelet counts reach ≥100 × 10⁹/L. The control group will not receive rh-TPO or any thrombopoietin receptor agonist (TPO-RA) therapy. Supportive care including transfusions and growth factors (G-CSF, ESA) is allowed in both groups.

The primary endpoint is the cumulative platelet engraftment rate by day +21 post-transplant, defined as sustained platelet counts > 20 × 10⁹/L for at least 7 consecutive days without transfusion. Secondary endpoints include median time to platelet engraftment, median time to achieve platelet counts ≥ 50 × 10⁹/L and ≥ 100 × 10⁹/L, total platelet transfusion volume, erythroid and neutrophil responses within 4 weeks, and overall hematopoietic recovery. Safety endpoints include the incidence of adverse events, thromboembolic events, and treatment-related serious adverse events.

The study aims to determine whether early administration of Romiplostim N01 can accelerate platelet recovery and reduce bleeding risk in patients undergoing haplo-HSCT, thereby improving post-transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients with malignant hematologic diseases scheduled to undergo haploidentical allogeneic hematopoietic stem cell transplantation (haplo-HSCT) Age ≥18 years, male or female. ECOG performance status 0-1. Estimated life expectancy >6 months. Adequate renal function, defined as:serum creatinine ≤1.5 × upper limit of normal (ULN);Blood urea nitrogen (BUN) ≤1.5 × ULN.

Adequate hepatic function, defined as:Alanine aminotransferase (ALT) ≤2 × ULN.Aspartate aminotransferase (AST) ≤2 × ULN.Total bilirubin ≤1.5 × ULN.

Ability to understand and sign informed consent, and willingness to comply with all study requirements.

Exclusion Criteria:

Uncontrolled active infection or other active malignancy that could interfere with study participation.

Severe cardiovascular disease, including:New York Heart Association (NYHA) Class III-IV heart failure;Uncontrolled hypertension or hypotension;History of or high risk for thromboembolic events.

Receiving anticoagulation therapy for thrombotic events. Known hypersensitivity to romiplostim or similar agents. Use of rh-TPO or any thrombopoietin receptor agonist (TPO-RA) within 30 days prior to enrollment.

Participation in another interventional clinical study within 30 days prior to enrollment.

Any other condition that, in the investigator's judgment, makes the patient unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative Platelet Engraftment Rate by Day +21 after Haploidentical HSCT | Within 21 days after transplantation
  Platelet engraftment is defined as achieving a sustained platelet count >20 × 10⁹/L for at least 7 consecutive days without platelet transfusion. The cumulative engraftment rate by day +21 post-transplant will be compared between the Romiplostim N01 treatment arm and the standard care control arm.

SECONDARY OUTCOMES:
Time to Platelet Engraftment | Up to 60 days after transplantation
  The number of days from transplantation to the first of 7 consecutive days with a platelet count >20 × 10⁹/L without transfusion support.
Proportion of Patients Achieving Platelet Counts ≥50 × 10⁹/L and ≥100 × 10⁹/L | Up to 60 days after transplantation
Median Time to Achieve Platelet Count ≥100 × 10⁹/L during the 4-Week Treatment Period | Within 4 weeks after initiation of Romiplostim N01 treatment
Total Platelet Transfusion Volume | Up to 60 days after transplantation
Proportion of Participants with Erythroid Response during the 4-Week Treatment Period | Within 4 weeks after initiation of Romiplostim N01 treatment
Proportion of Participants with Neutrophil Response during the 4-Week Treatment Period | Within 4 weeks after initiation of Romiplostim N01 treatment

OTHER OUTCOMES:
Incidence of Thrombotic or Thromboembolic Events | Within 4 weeks after initiation of Romiplostim N01 treatment
Incidence of Treatment-Related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) | From initiation of treatment up to 100 days after transplantation
Incidence of Adverse Events (AEs) | From initiation of Romiplostim N01 to 100 days after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, China